CLINICAL TRIAL: NCT00693992
Title: Randomized, Phase III, Double-Blind Placebo-Controlled Trial of Sunitinib (NSC #736511) as Maintenance Therapy in Non-progressing Patients Following an Initial Four Cycles of Platinum-Based Combination Chemotherapy in Advanced, Stage IIIB / IV Non-small Cell Lung Cancer
Brief Title: Sunitinib Malate as Maintenance Therapy in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer Previously Treated With Combination Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2009-00469; NCI-2009-00469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000597649; CALGB 30607 (Other: Alliance for Clinical Trials in Oncology); CALGB-30607 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH); NCT01647087 (obsolete NCT alias)
Record Dates: First submitted 2008-06-06; First posted 2008-06-09 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (sunitinib malate) (Experimental): Patients receive sunitinib malate 37.5 mg PO once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Sunitinib Malate
- Arm II (placebo) (Placebo Comparator): Patients receive placebo 37.5 mg PO once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
  Arms: Arm I (sunitinib malate)

SUMMARY:
This randomized phase III trial studies sunitinib malate to see how well it works when given as maintenance therapy (meaning it is approved for treatment after chemotherapy) in patients with stage IIIB-IV non-small cell lung cancer who have responded to prior treatment with combination chemotherapy. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking the growth of new blood vessels necessary for tumor growth. It is not yet known whether sunitinib malate is effective in helping tumors continue to shrink or stop growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of sunitinib (sunitinib malate) compared to placebo on progression-free survival (PFS) in advanced non-small cell lung cancer (NSCLC) patients who have had either stable or responding disease over the course of their initial 4 cycles of platinum-based therapy.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of sunitinib compared to placebo in the maintenance setting.

II. To evaluate the additional response rate as a result of sunitinib in this setting.

III. To assess the impact of sunitinib on overall survival compared to the placebo arm.

IV. To assess the impact of sunitinib on delaying the time to deterioration in quality of life and symptom progression compared to placebo using the European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30) and Lung Cancer Module (LC13).

V. To assess vascular endothelial growth factor (VEGF) haplotypes in advanced non-small cell lung cancer and sunitinib maintenance.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 1 year, and then periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic documentation of primary non-small cell lung cancer
* Stage IIIB or IV disease patients who are not candidates for combined modality therapy (chemoradiotherapy)
* No evidence of symptomatic or untreated brain metastases, spinal cord compression, or carcinomatous meningitis; patients with central nervous system (CNS) metastases must be asymptomatic, must have received definitive therapy (>= 6 weeks since resection or >= 2 weeks since radiotherapy) for brain metastases, and be off steroids or on a stable dose for 2 weeks prior to registration
* No cavitary lesions
* Patients must have received one chemotherapy regimen for stage IIIB or IV NSCLC; the regimen must include four cycles of platinum-based doublet chemotherapy with or without bevacizumab (bevacizumab may not be given beyond the fourth cycle of chemotherapy); patients must have achieved a complete response, partial response, or stable disease to first-line chemotherapy and have no evidence of disease progression; patients will be registered 3-5 weeks following day 1 of cycle 4 of prior therapy
* No prior adjuvant chemotherapy for stage I-III resected NSCLC or combined modality therapy for stage III NSCLC
* No other primary therapy (including experimental therapy) for NSCLC; palliative radiation therapy must have been completed at least one week before planned start of protocol therapy
* Patients must have measurable or non-measurable disease

  * Measurable disease: lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan
  * Non-measurable disease: all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions; lesions that are considered non-measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Non-pregnant and non-nursing
* No ongoing cardiac dysrhythmias, atrial fibrillation, or history of corrected QT (QTc) interval >= 500 msec (within 2 years prior to registration); the use of agents with proarrhythmic potential (e.g., quinidine, procainamide, disopyramide, sotalol, probucol, haloperidol, risperidone, indapamide, flecainide) is not recommended while on protocol therapy
* Patients with class I New York Heart Association (NYHA) heart failure are eligible; patients with a history of class II NYHA heart failure are eligible, provided they meet at least one of the following criteria:

  * Patients with a history of class II heart failure who are asymptomatic on treatment
  * Patients with prior anthracycline exposure
  * Patients who have received central thoracic radiation that included the heart in the radiotherapy port
* Patients with a history of class III or IV NYHA heart failure within 12 months prior to registration are not eligible
* No myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft or stenting, cerebrovascular accident or transient ischemic attack within the last year
* Patients with hypertension that cannot be controlled by medications (> 150/100 mmHg despite optimal medical therapy) are not eligible
* Patients who require use of therapeutic anticoagulation for thromboembolic disease are not eligible; Note: low doses of coumadin (up to 2 mg daily) are permitted for prophylaxis of thrombosis
* No history of venous thrombosis, pulmonary embolism, or hypercoagulopathy syndrome
* No history of pulmonary hemorrhage, bleeding diathesis, or evidence of hemoptysis; patients with blood-tinged or blood-streaked sputum will be permitted on study if the hemoptysis amounts to less than 5 ml of blood per episode and less than 10 ml of blood per 24-hour period in the best estimate of the investigator
* Patients with a history of hypothyroidism are eligible, provided they are currently euthyroid
* None of the following within 28 days of beginning treatment: abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, serious or non-healing wound, ulcer, or bone fracture
* The following inhibitors of cytochrome P450 3A4 (CYP3A4) are prohibited within 7 days before beginning and during treatment with sunitinib: azole antifungals (ketoconazole, itraconazole), diltiazem, clarithromycin, erythromycin, verapamil, delavirdine, and human immunodeficiency virus [HIV] protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir); the following inducers of CYP3A4 are prohibited within 12 days before beginning and during treatment with sunitinib: rifampin, rifabutin, carbamazepine, phenobarbital, phenytoin, St. John?s Wort, efavirenz, tipranavir; other inhibitors and inducers of CYP3A4 may be used if necessary, but their use is discouraged
* Patients unable to take oral medication are not eligible
* Granulocytes >= 1,500/mcl
* Platelet count >= 100,000/mcl
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)=< 2.5 x ULN; patients with liver metastases may have AST and ALT =< 5 x ULN; all other patients will have AST and ALT =< 2.5 x ULN
* Creatinine =< 1.5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-06-15 (Actual); Primary Completion 2013-11-08 (Actual); Study Completion 2015-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Socinski, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (484):
- United States (484):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Providence Hospital, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Feather River Cancer Center, Chico, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Saint Helena Hospital, St. Helena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - AMG Oncology - Naperville, Naperville, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Veterans Administration Medical Center-Baltimore, Baltimore, Maryland
  - MedStar Harbor Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Beverly Hospital, Beverly, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Nash General Hospital, Rocky Mount, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Coastal Cancer Center-Myrtle Beach, Myrtle Beach, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Baggstrom MQ, Socinski MA, Wang XF, Gu L, Stinchcombe TE, Edelman MJ, Baker S Jr, Feliciano J, Novotny P, Hahn O, Crawford JA, Vokes EE. Maintenance Sunitinib following Initial Platinum-Based Combination Chemotherapy in Advanced-Stage IIIB/IV Non-Small Cell Lung Cancer: A Randomized, Double-Blind, Placebo-Controlled Phase III Study-CALGB 30607 (Alliance). J Thorac Oncol. 2017 May;12(5):843-849. doi: 10.1016/j.jtho.2017.01.022. Epub 2017 Feb 1. PMID 28161554
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Started | 106 | 104
Completed | 106 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo) | Total
Number analyzed (Participants) | 106 | 104 | 210
Age, Continuous [Median (Full Range); unit: years] | 65 [25 to 84] | 67 [44 to 89] | 66 [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 44 | 93
  Male | 57 | 60 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 13 | 31
  White | 87 | 85 | 172
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 106 | 104 | 210

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) was defined as the time from randomization until disease progression or death, whichever occurs first. The median PFS with 95% CI was estimated using the Kaplan-Meier method. Progression is defined as in the primary outcome measure.
Time Frame: Time from randomization to disease progression and death of any cause, whichever comes first (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Number analyzed (Participants) | 106 | 104
months | 4.3 [3.2 to 4.9] | 2.6 [1.8 to 3.0]
Statistical Analysis 1: Comparison: Arm I (Sunitinib Malate) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.0006, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.47 to 0.82]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from patient randomization to death from any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Time from randomization to death (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Number analyzed (Participants) | 106 | 104
months | 11.7 [9.9 to 14.0] | 12.1 [9.8 to 15.3]
Statistical Analysis 1: Comparison: Arm I (Sunitinib Malate) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.89, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.73 to 1.31]

3. Secondary Outcome: Response Rate (RR)
Description: The percentage of patients who respond (completely or partially) to each combination regimen will be estimated. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions.
Time Frame: Duration of treatment (up to 5 years)
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Number analyzed (Participants) | 106 | 104
percentage of participants | 11 | 5

4. Secondary Outcome: Percentage of Deterioration in QOL at 3 Months Using the EORTC QLQ-C30 Global Health Subscale
Description: The percentage of patients with at least a 10% drop in the EORTC-QLQ-C30 Global Health Subscale score from baseline to 3-months. The difference between groups will be tested using Fisher's exact test.
Time Frame: At 3 months
Population: Patients who completed the EORTC-QLQ-C30 Global Health Subscale at baseline and 3 months were included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Number analyzed (Participants) | 80 | 83
percentage of patients | 55.8 | 28.6
Statistical Analysis 1: Comparison: Arm I (Sunitinib Malate) vs Arm II (Placebo); Test type: Superiority; p = 0.0061, Fisher Exact

5. Secondary Outcome: Percentage of Deterioration in Symptom Progression at 3 Months Using the EORTC LC13 Dyspnea Subscale
Description: The percentage of patients with at least a 10% drop in the EORTC LC13 Dyspnea Subscale score from baseline to 3-months. The difference between groups will be tested using Fisher's exact test.
Time Frame: At 3 months
Population: Patients who completed the EORTC LC13 Dyspnea Subscale at baseline and 3 months were included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Number analyzed (Participants) | 83 | 85
percentage of patients | 31.5 | 29.3
Statistical Analysis 1: Comparison: Arm I (Sunitinib Malate) vs Arm II (Placebo); Test type: Superiority; p = 0.8393, Fisher Exact

6. Secondary Outcome: Grade and Type of Toxicity as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Grade 3 or 4 adverse events which affected more than 5% of participants are summarized by arm.
Time Frame: Duration of study (up to 5 years)
Population: 189 participants were evaluable for adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Number analyzed (Participants) | 97 | 92
percentage of participants
  Fatigue | 26 | 0
  Thrombocytopenia | 12 | 0
  Hypertension | 12 | 0
  Rash | 11 | 0
  Mucositis | 11 | 0
  Neutropenia | 7 | 0
  Anemia | 6 | 0

7. Other Pre Specified Outcome: VEGF Levels and Correlation With Clinical Outcomes, Including RR, PFS, and OS
Time Frame: Up to 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 189 participants were evaluable for adverse events.
Arm/Group | Arm I (Sunitinib Malate) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 33/97 | 14/92
Other Adverse Events (participants affected / at risk) | 87/97 | 85/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sunitinib Malate) (N=97) | Arm II (Placebo) (N=92)
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 (11) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 5 (5)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 26 (34) | 8 (9)
Fever (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Electrocardiogram QTc interval prolonged (Investigations) | 2 (2) | 0 (0)
Leukocyte count decreased (Investigations) | 3 (4) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 0 (0)
Platelet count decreased (Investigations) | 9 (11) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 12 (13) | 2 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 7 (8) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sunitinib Malate) (N=97) | Arm II (Placebo) (N=92)
Hemoglobin decreased (Blood and lymphatic system disorders) | 9 (28) | 3 (6)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (9)
Left ventricular failure (Cardiac disorders) | 1 (1) | 2 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (11) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 44 (112) | 15 (37)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mouth necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 34 (71) | 7 (14)
Nausea (Gastrointestinal disorders) | 37 (73) | 20 (42)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (10) | 1 (1)
Chest pain (General disorders) | 3 (4) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 4 (13)
Fatigue (General disorders) | 69 (218) | 67 (204)
Fever (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (3) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury to superior vena cava (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 2 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (12) | 3 (15)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1) | 2 (4)
Leukocyte count decreased (Investigations) | 7 (23) | 2 (9)
Lipase increased (Investigations) | 1 (1) | 2 (4)
Lymphocyte count decreased (Investigations) | 3 (6) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (23) | 1 (1)
Platelet count decreased (Investigations) | 13 (24) | 1 (2)
Weight loss (Investigations) | 4 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 32 (83) | 19 (34)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (2) | 7 (31)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (12) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (7) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (2) | 2 (7)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (6)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (3) | 1 (7)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (8) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 6 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Accessory nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (8) | 1 (1)
Headache (Nervous system disorders) | 15 (27) | 12 (26)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (15) | 5 (7)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 28 (83) | 8 (14)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 9 (21) | 0 (0)
Hemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 29 (81) | 13 (41)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less